CLINICAL TRIAL: NCT06844656
Title: Understanding the Increased Risk of Atrial Fibrillation in Athletes: a Case-control Study
Acronym: AFLETES-ECG
Status: Not yet recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 1001
Record Dates: First submitted 2025-01-27; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Athletes; Sport; Physical Activity; Exercise; Arrhythmias
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, buffycoat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AF Athletes: Athletes with atrial fibrillation.
- Non-AF Athletes: Athletes without atrial fibrillation.

SUMMARY:
Exercise is beneficial to heart health, however, there appears to be a 'U' shaped relationship where too much exercise may increase the risk of an irregular heart rhythm, called atrial fibrillation. Endurance athletes may have up to a 2.5-fold higher risk of developing atrial fibrillation than non-athletic controls.

The mechanisms behind this increased risk of atrial fibrillation are not the well understood. It is thought to be a mixture of enlarged heart chambers, low resting heart rate, genetic predisposition and possibly scarring in the heart. In this study, the investigators will investigate the electrical activity changes in the heart, using a high-quality electrocardiogram (ECG) and relate this to changes in the heart size measured by ultrasound and MRI. Cardiopulmonary exercise testing will determine fitness (V̇O2 max) and assess the heart's electrical activity during exercise.

This will be a case-control study where athletes with and without atrial fibrillation will be recruited. The investigators hope the results of this study can improve our understanding of atrial fibrillation in athletes by associating atrial fibrillation with structural and electrical differences which may aid the prediction of future atrial fibrillation development and help guide more athlete-specific treatment pathways.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of enrolment, male and female.
* History of atrial fibrillation confirmed on ECG - either paroxysmal or persistent.
* Competitive athlete. Defined as:

  1. Competed in endurance sports with a total cumulative moderate to high intensity of > 1500 hours.
  2. Have participated in at least one competitive event in the last 10 years.

Exclusion Criteria:

* Permanent atrial fibrillation.
* History of pre-existing cardiovascular disease :

  1. Atherosclerotic disease: previous myocardial infarction, symptomatic coronary artery disease or Peripheral peripheral arterial disease
  2. Left ventricular systolic dysfunction (EF < 45%)
  3. Heart muscle disease: cardiomyopathies, Infiltrative diseases of the heart
  4. Complex Congenital heart disease
  5. Moderate or severe valvular disease
  6. Uncontrolled hypertension (>180/100mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endurance athletes with and without atrial fibrillation from across the United Kingdom. Recruitment through social media, sports clubs, and word of mouth.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
High-resolution ECG | At study visit
  Using high quality ECG, assess whether subtle differences can be detected in athletes with AF, compared to athletes without AF, and whether machine learning could predict new-onset AF.
  Detection of subtle differences in p wave parameters (duration, amplitude, dispersion, PTFV1) in athletes with AF compared to athletes without AF. AUC, specificity and sensitivity.

SECONDARY OUTCOMES:
AI classification and prediction | At study visit
  Assess the accuracy of using machine learning to identify athletes with AF using ECG data.
  AUC, specificity and sensitivity of machine learning identification of AF.
72hr heart rate monitoring | At study visit
  Compare autonomic tone via heart rate variability from 72-hour continuous ECG monitoring in athletes with and without AF.
  Analysis of RR intervals from heart rate variability.
Electronic stethoscope recording | At study visit
  Compare the heart sounds using electronic stethoscope in athletes with and without AF.
  S1 and S2 sounds of heart valves.
Cardiac imaging | At study visit
  Left ventricular mass
Cardiac imaging | At study visit
  Left ventricular volume
Cardiac imaging | At study visit
  Strain rate
Cardiac imaging | At study visit
  Myocardial perfusion reserve
Cardiac imaging | At study visit
  Myocardial interstitial fibrosis
Cardiac imaging | At study visit
  Left atrial mass
Cardiac imaging | At study visit
  Left atrial volume
Cardiac imaging | At study visit
  Vascular stiffness
Cardiac imaging | At study visit
  Left ventricular filling pressure
Cardiac imaging | At study visit
  Tissue Doppler velocity
Cardiopulmonary exercise testing | At study visit
  Peak VO2
Cardiopulmonary exercise testing | At study visit
  Exercising p wave duration
Cardiopulmonary exercise testing | At study visit
  Exercising p wave amplitude
Cardiopulmonary exercise testing | At study visit
  Exercising p wave dispersion
Cardiopulmonary exercise testing | At study visit
  Exercising p wave PTFV1
Cardiac motion recording | At study visit
  Cardiac angular velocity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiovascular Sciences. University of Leicester. Glenfield Hospital., Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant identifiable data will not be shared. Imaging scans anonymised may be shared with future potential collaborators.